CLINICAL TRIAL: NCT00005579
Title: Phase II Trial of Dolastin 10 in Indolent Lymphoma and Chronic Lymphocytic Leukemia
Brief Title: Dolastatin 10 in Treating Patients With Indolent Lymphoma, Waldenstrom's Macroglobulinemia, or Chronic Lymphocytic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Vermont (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: VCC-9802; CDR0000066360 (Registry Identifier: PDQ (Physician Data Query)); NCI-T98-0007
Record Dates: First submitted 2000-05-02; First posted 2003-01-27 (Estimated); Last update posted 2013-06-26 (Estimated); Status verified 2002-11

CONDITIONS: Leukemia; Lymphoma
Keywords: Waldenström macroglobulinemia; stage I chronic lymphocytic leukemia; stage II chronic lymphocytic leukemia; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia; refractory chronic lymphocytic leukemia; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV adult diffuse small cleaved cell lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent small lymphocytic lymphoma; stage III small lymphocytic lymphoma; stage IV small lymphocytic lymphoma
MeSH Terms: conditions — Leukemia; Lymphoma; Waldenstrom Macroglobulinemia; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Follicular; Lymphoma, Non-Hodgkin | interventions — dolastatin 10

INTERVENTIONS:
Drug: dolastatin 10

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of dolastatin 10 in treating patients with indolent lymphoma, Waldenstrom's macroglobulinemia, or chronic lymphocytic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Estimate the efficacy of dolastatin 10 in patients with indolent lymphoma, Waldenstrom's macroglobulinemia, or chronic lymphocytic leukemia.
* Evaluate the qualitative and quantitative toxicities of dolastatin 10 in this patient population.
* Investigate the mechanism of action of dolastatin 10 in regards to apoptosis and effects of microtubules.

OUTLINE: This is an open-label, multicenter study. Patients are stratified by disease (chronic lymphocytic leukemia vs indolent lymphoma vs Waldenstrom's macroglobulinemia).

All patients receive dolastatin 10 IV bolus every 3 weeks. Patients continue treatment until disease progression, unacceptable toxicity, or patient's withdrawal from the study.

PROJECTED ACCRUAL: A maximum of 74 patients will be accrued for this study over 15 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologic or cytologic diagnosis of indolent lymphoma as defined by International Working Formulation categories A-C or diagnosis of Waldenstrom's macroglobulinemia, or chronic lymphocytic leukemia
* Lymphoma must be stage III, IV, or recurrent (no primary CNS lymphoma or lymphomatous meningitis)
* Waldenstrom's macroglobulinemia must have at least one of the following:

  * IGM greater than 3,000 mg/dL
  * Hemoglobin less than 10.0 g/dL
  * Bone marrow involvement greater than 30% lymphocytes
  * At least 2 cm lymphadenopathy
  * Serum viscosity greater than 3.0
* Chronic lymphocytic leukemia must be intermediate or high risk stages I-IV and have progressed on fludarabine therapy unless patient cannot tolerate fludarabine

  * Intermediate risk group must have at least one indication of active disease:

    * Presence of any one of the disease related B symptoms: 10% or more loss of body weight over the preceding 6 month period, extreme fatigue, fever above 100 degrees F without evidence of infection, or night sweats
    * Massive (greater than 6 cm below left costal margin) or progressive splenomegaly
    * Massive (greater than 10 cm in longest diameter) or progressive lymphadenopathy
    * Progressive lymphocytosis with an increase of 50% over a 2 month period or anticipated doubling time of less than 12 months
    * Evidence of progressive marrow failure as manifested by the development or worsening of anemia and/or thrombocytopenia
    * Autoimmune anemia and/or thrombocytopenia poorly responsive to corticosteroid therapy
* Intolerance, relapse, or failure following prior fludarabine allowed
* Measurable or evaluable disease
* No untreated immediate life threatening tumor complications

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* CALGB 0-2

Life expectancy:

* Not specified

Hematopoietic:

* See Disease Characteristics
* WBC at least 4,000/mm^3*
* Absolute granulocyte count at least 1,500/mm^3*
* Platelet count at least 100,000/mm^3*
* Hemoglobin at least 9 g/dL* NOTE: *Unless documented bone marrow involvement

Hepatic:

* Bilirubin no greater than 1.5 mg/dL
* SGOT no greater than 2.5 times upper limit of normal

Renal:

* Creatinine no greater than 1.5 mg/dL OR
* Creatinine clearance at least 60 mL/min

Other:

* No prior malignancy except adequately treated basal or squamous cell skin cancer, carcinoma in situ of the cervix, well differentiated stage IA prostate cancer, or any other cancer from which the patient has been disease free for five years
* Not pregnant or nursing
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior autologous bone marrow or stem cell transplantation

Chemotherapy:

* See Disease Characteristics
* No more than 2 prior systemic regimens for treatment of lymphoma
* No chemotherapy for treatment of any other prior malignancy
* At least 4 weeks since chemotherapy and recovered
* Prior fludarabine therapy allowed

Endocrine therapy:

* See Disease Characteristics

Radiotherapy:

* Prior radiotherapy allowed (index lesion cannot be within prior radiotherapy field)

Surgery:

* Recovered from prior surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1998-06; Study Completion 2003-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven M. Grunberg, MD, Study Chair — University of Vermont
Locations (4):
- United States (4):
  - Marlene and Stewart Greenebaum Cancer Center, University of Maryland, Baltimore, Maryland
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - Vermont Cancer Center, Burlington, Vermont